CLINICAL TRIAL: NCT06776094
Title: The Significance of Physical Activity for Insulin Signaling Dynamics and Insulin Sensitivity
Brief Title: Physical Activity and Insulin Sensitivity Dynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jorgen FP Wojtaszewski, Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TEMPO
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Insulin Sensitivity
Keywords: Exercise; Muscle insulin sensitivity; Muscle glucose uptake; GLUT4; Phosphoproteomics
MeSH Terms: conditions — Insulin Resistance; Motor Activity | interventions — Insulin Infusion Systems; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-exercise insulin sensitivity (Experimental): Young healthy males will perform a single bout of knee-extensor exercise and insulin action is investigated 4 hours after cessation of exercise. Insulin action towards muscle glucose uptake will be investigated during a 120 min euglycemic hyperinsulinemic clamp.
  Interventions: Other: One-legged-knee extensor exercise; Procedure: Insulin infusion; Procedure: Muscle Biopsy Medication: Lidocaine; Other: Exercise

INTERVENTIONS:
Other: One-legged-knee extensor exercise — 1 hour of one-legged-knee-extensor exercise followed by 4 hours of rest
Procedure: Insulin infusion — The hyperinsulinemic-euglycemic clamp is a well-established and recognized method for determining glucose uptake at a specific insulin infusion rate. It is a technique with which we have 25 years of uncomplicated experience. During the clamp, insulin (human recombinant insulin) is infused (1.42 mU/kg/min) into an arm vein (antecubital vein), while glucose (20% solution) is administered in an amount adjusted to maintain blood glucose (plasma glucose concentration) at basal levels.
  The amount of insulin administered raises the participant's plasma insulin concentration (blood concentration) to approximately 100 μU/mL, which is considered within the physiological range. Blood samples are collected and analyzed continuously for glucose content, allowing for the determination of glucose uptake at the whole-body level and across the legs.
  Later, these blood samples will also be analyzed for relevant metabolites and proteins, including insulin, to assess the metabolism of these substances.
Procedure: Muscle Biopsy Medication: Lidocaine — During supine rest, the skin on the outer thigh, approximately 15 cm above the knee, is disinfected with chlorhexidine alcohol. Subsequently, 3-4 mL of local anesthetic (lidocaine 20 mg/mL) is administered into the skin, subcutaneous tissue, and the upper portion of the muscle using a very thin needle. A pinprick test is performed after a few minutes to ensure the anesthetic is effective.
  A small incision is then made in the skin and subcutaneous tissue to allow the biopsy needle to pass through to the muscle. Using the biopsy needle, a small sample of muscle tissue (approximately 150 mg) is collected. This may cause some discomfort but is very brief (~1-2 seconds). The needle is removed, a sterile dressing is applied, and the participant can leave the facility after completing the study.
  The biopsy may result in mild muscle soreness for 2-3 days, similar to a minor muscle bruise. Regular physical activities can be resumed after the biopsy. However, it is advised to avoid swimming.
Other: Exercise — The participants' maximal oxygen uptake is determined through a test on a cycle ergometer before the start of the experiment. The test begins with a 20-minute warm-up at two different low workloads, after which the workload is gradually increased until the predetermined cadence can no longer be maintained, or the participant indicates exhaustion. During the test, the participant's exhaled air is collected. After completing the warm-up, it typically takes between 4 and 7 minutes to complete the test.

SUMMARY:
The study investigates the role of one single bout of exercise in mediating enhancement of muscle insulin sensitivity following a single bout of exercise. Furthermore, the study is aiming to elucidate the temporal development in insulin signaling, at the early timepoints of insulin stimulation that may be responsible for the enhanced muscle insulin sensitivity.

This will be investigated in young healthy males subjected to a one-legged knee-extensor exercise followed by a hyperinsulinemic-euglycemic clamp, a setup known to enhance muscle insulin sensitivity.

DETAILED DESCRIPTION:
The participant arrives fasting at 8:00 AM, having abstained from alcohol, nicotine, and caffeine for the past 24 hours and refrained from strenuous physical activity for the past 48 hours. The participants are then subjected to a one-legged knee extension exercise performed by the participant from 9:00 AM to 10:00 AM.

Groin catheters are inserted into the femoral artery and vein using ultrasound guidance and sterile technique

Two hours after the completion of the exercise, a catheter is inserted into an arm vein (antecubital vein) and groin catheters are inserted into the femoral artery and vein using ultrasound guidance and sterile technique. Four hours after the exercise ends, a hyperinsulinemic-euglycemic clamp is commenced. The clamp begins with a bolus injection of insulin, followed by a continuous infusion. Glucose is infused concurrently to maintain constant blood glucose levels.

Throughout the procedure, blood samples are collected every 5 minutes from the femoral catheters, and blood flow is measured using ultrasound Doppler. Muscle biopsies from the vastus lateralis of both legs are taken before the clamp starts and at 3, 6, 10, and 20 minutes after the clamp's initiation. Following the 20-minute mark, the clamp continues until steady-state is achieved to determine tissue-specific and whole-body insulin sensitivity.

Over the course of the experiment, a total of 10 muscle biopsies and approximately 150 mL of blood are collected. The experimental part of the study is expected to conclude by 4:30 PM. Participants are provided with food and beverages and observed for 1 hour before being allowed to leave the research laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (no known diseases)
* No use of medication
* Non-smokers
* Male
* Aged 22-35 years
* Fitness level (VO2max, i.e., maximal oxygen uptake) between 30-50 mL O2/min/kg
* BMI between 28 and 35

Exclusion Criteria:

* Women
* Failure to meet all inclusion criteria
* Physical activity level (e.g., running, cycling, fitness, etc.) exceeding 6 hours per week
* Acute illness within 2 weeks prior to the study days
* Use of recreational drugs within 2 weeks prior to the study days

Ages: 22 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Insulin stimulated muscle glucose uptake | Through study completion, approx. 1 year.
  Muscle glucose uptake during insulin stimulation in recovery from exercise (insulin sensitivity) will be determined based on Fick's principle. Thus, femoral arterio-venous difference (av difference) in blood glucose concentration will be multiplied by femoral arterial leg blood flow.

SECONDARY OUTCOMES:
Posttranslational modification of proteins in muscle biopsies | 3 years
  The obtained muscle samples will be subjected to mass spectrometry-based phosphoproteomic analysis. This measurement shows posttranslational modification that regulates protein function and will reveal the signalling network underlying the interventions studied. Unit of measure is log2-transformed arbitrary units

OTHER OUTCOMES:
Imaging of transport protein | 1 year
  The obtained muscle samples will be subjected to a microscopy method to validate the spatial distribution and re distribution following insulin stimulation.
Maximum oxygen uptake | Through study completion, approx. 1 year.
  The participants' maximal oxygen uptake is determined through a test on a cycle ergometer before the start of the experiment. The test begins with a 20-minute warm-up at two different low workloads, after which the workload is gradually increased until the predetermined cadence can no longer be maintained, or the participant indicates exhaustion. During the test, the participant's exhaled air is collected. After completing the warm-up, it typically takes between 4 and 7 minutes to complete the test.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen FP Wojtaszewski, Prodessor, Principal Investigator — Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- University of Copenhagen, August Krogh Section for Human and Molecular Physiology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No